CLINICAL TRIAL: NCT01587326
Title: The Effects of Escitalopram on Cytokines in Depressive Patients
Brief Title: The Effects of Escitalopram on Cytokines
Acronym: BAFH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beitou Armed Forces Hospital, Taipei, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BAFH-101-05; BAFH (Other: Civilian Administration Division)
Record Dates: First submitted 2012-04-26; First posted 2012-04-30 (Estimated); Last update posted 2012-05-15 (Estimated); Status verified 2012-05

CONDITIONS: Depression
Keywords: cytokine, depression, escitalopram
MeSH Terms: conditions — Depression | interventions — Escitalopram

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Escitalopram (Experimental): Escitalopram 10 mg/d to 20 mg/d
  Interventions: Drug: Escitalopram

INTERVENTIONS:
Drug: Escitalopram — escitalopram 10 mg/d to 20 mg/d
  Other Names: Lexapro

SUMMARY:
The association of cytokines with escitalopram has not been investigated in patients with major depressive disorder (MDD). Hence, the investigators will examine this association.

DETAILED DESCRIPTION:
In addition to serotonin, inflammatory process has been suggested in the development of major depressive disorder (MDD) and in its associated treatment. Escitalopram is an antidepressant that has been widely used in patients with MDD because of the promising results. The association of cytokines with escitalopram has not been investigated in patients with MDD. Hence, the investigators will examine this association.

ELIGIBILITY:
Inclusion Criteria:

1. DSM-IV-defined Major depressive disorder, single episode
2. Age 20-65
3. Drug-naive
4. Hamilton Depression Rating Scale exceeding 14 scores

Exclusion Criteria:

1. Major medical disorders
2. Substance use
3. Pregnant
4. Allergy to escitalopram

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2012-04; Primary Completion 2013-04 (Estimated); Study Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
The changes in cytokines | Week 0, Week 4
  Hamilton Depression Rating Scale, IL-1β, IL-2, IL-4, IL-5, IL-6, IL-7, IL-8, IL-10, IL-12, IL-13, IL-17A, G-CSF, GM-CSF, IFN-γ, MCP-1, MIP-1β, TNF-α

SECONDARY OUTCOMES:
The changes in Hamilton Depression Rating Scale | week 0, week 4
  Hamilton Depression Rating Scale, IL-1β, IL-2, IL-4, IL-5, IL-6, IL-7, IL-8, IL-10, IL-12, IL-13, IL-17A, G-CSF, GM-CSF, IFN-γ, MCP-1, MIP-1β, TNF-α

CONTACTS AND LOCATIONS:
Overall Officials: Peishen Ho, M.D., Study Chair — Beitou Armed Forces Hospital
Locations (1):
- Beitou Armed Forces Hospital, Taipei, Taiwan